CLINICAL TRIAL: NCT04236570
Title: Evaluation of Endogenous Pain Modulation Mechanisms With Transcutaneous Electrical Nerve Stimulation (TENS)
Brief Title: Evaluation of Endogenous Pain Modulation Mechanisms With Transcutaneous Electrical Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019-3022
Record Dates: First submitted 2020-01-07; First posted 2020-01-22 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Chronic Pain
Keywords: Excitatory mechanisms; Inhibitory mechanisms; Thermode(hot plate); Cold water bath; Transcutaneous electrical nerve stimulation (TENS)
MeSH Terms: conditions — Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will attended two experimental sessions at the Research Center on Aging of the Centre Intégré Universitaire de Santé et de Services Sociaux de l'Estrie, Sherbrooke, during which the efficacy of their excitatory and inhibitory mechanisms was assessed. In one session, this assessment was done using TENS protocol; in the other, using a standardized protocol (thermode and cold water bath). Session order was randomized between participants (randomization by block of 4 stratified by sex, using a random number table). The two sessions were separated by 24 to 72 hours and lasted approximately one hour each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain tests with the standardized protocol (Other): This arm will consisted of pain tests using the standardized protocol (thermode(hot plate) and cold water bath)). The investigators will used the modified CPM testing procedure consisting of stimulus test (TS) administered before and after a conditioning stimulus (CS). For the standardized protocol, the TS will consisted of a noxius heat stimulus generated by a thermode (hot plate), applied for two minutes on the non-dominant anterior forearm. The CS will consisted of a cold pressor test (CT), wherein participants immersed their dominant forearm in a cold water bath for two minutes.
  Interventions: Device: Thermode(hot plate) and cold water bath
- Pain tests with the TENS protocol (Other): This arm will consisted of pain tests using the TENS protocol. The investigators will used the modified CPM testing procedure consisting of stimulus test (TS) administered before and after a conditioning stimulus (CS). For the TENS protocol, the TS will consisted of a noxius electrical stimulus generated by TENS, applied for 5 seconds on the non-dominant knee at a frequency of 1 Hz and 5 Hz. The CS will consisted of a noxius electrical stimulus generated by TENS' applied for 120 seconds on the non dominant knee and ankle at a frequency of 2 Hz
  Interventions: Device: TENS(transcutaneous electrical nerve stimulation)

INTERVENTIONS:
Device: Thermode(hot plate) and cold water bath — Standardized protocol will consisted of stimulus test (TS) generated by thermode and conditioning stimulus (CS) using cold water bath.
  Arms: Pain tests with the standardized protocol
Device: TENS(transcutaneous electrical nerve stimulation) — TENS protocol will consisted of test stimulus (TS) and conditioning stimulus (CS) both generated by TENS
  Arms: Pain tests with the TENS protocol

SUMMARY:
A number of chronic pain conditions are characterized by imbalances in excitatory and/or inhibitory mechanisms and these deficits appear correlated with the response to certain treatments. Evaluating these mechanisms among people who suffer from chronic pain could allow clinicians to adapt the treatment to each patient according to the deficits observed. To evaluate excitatory and inhibitory mechanisms, a thermode (hot plate) and a cold water bath can be used (standardized protocol). Unfortunately, these tools are expensive, time-consuming and require complex equipment and software. As such, it is not realistic for clinicians to use them for routine patient assessment. A potential alternative to study these mechanisms is TENS (transcutaneous electrical nerve stimulation). TENS is frequently used in rehabilitation and unlike thermode and cold water bath, is affordable, easy to use and requires very little time and equipment. The objective of this study are to determine if the TENS can replace the thermode and cold water bath (standardized protocol) for the evaluation of excitatory and inhibitory mechanisms. Also, to determine if there will be a correlation with the standardized protocol. 50 healthy participants between 18 and 60 years old will participate in this study. Each participant will attend two experimental sessions. In one of the two sessions, the evaluation will be done with the TENS; in the other session, the evaluation will be done with the standardized protocol (thermode and cold water bath).

DETAILED DESCRIPTION:
To evaluate excitatory and inhibitory mechanisms, the investigators will used the modified CPM testing procedure consisting of test stimulus (TS) administered before and after a conditioning stimulus (CS). For the standardized protocol, the TS will consisted of a noxius heat stimulus generated by a thermode (hot plate), applied for two minutes on the non-dominant anterior forearm. The CS will consisted of a cold pressor test (CT), wherein participants immersed their dominant forearm in a cold water bath for two minutes. For the TENS protocol, the TS will consisted of a noxius electrical stimulus generated by TENS, applied for 5 seconds on the non-dominant knee at a frequency of 1 Hz and 5 Hz. The CS will consisted of a noxius electrical stimulus generated by TENS' applied for 120 seconds on the non dominant knee and ankle at a frequency of 2 Hz.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18 and 60 years old (inclusive)

Exclusion Criteria:

* Chronic pain
* Neurological disorders
* Musculoskeletal disorders
* Depression
* Raynaud syndrome
* History of non-efficacy with TENS
* History of epilepsy
* Presence of a pacemaker or metal implants
* Antidepressant
* Anticonvulsant
* Analgesics
* Caffeine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate excitatory mechanisms, specifically temporal summation | This outcomes (excitatory pain mechanisms) will be evaluated at both sessions (V1 [day 0] and V2 [day 7])
  To evaluate excitatory mechanisms ,we will calculated if there is an increase of pain levels during the test stimulus (TS). Pain levels will be measured with a computerized visual analogue scale (CoVAS)
Evaluate inhibitory mechanisms, specifically conditioning pain modulation (CPM) | This outcome (mechanisms) will be evaluated at both sessions (V1 [day 0] and V2 [day 7])
  To evaluate inhibitory mechanisms ,we will calculated if there is an decrease of pain levels after the conditioning stimulus (CS). Pain levels will be measured with a computerized visual analogue scale (CoVAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No